CLINICAL TRIAL: NCT07347678
Title: A Phase 1a, Randomized, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RN5681 in Healthy Volunteers
Brief Title: Phase 1a Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RN5681 in Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ikaria Bioscience Pty Ltd (Industry)
Collaborators: Shanghai Rona Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RN5681-101
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-01

CONDITIONS: High Cholesterol
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RN5681 (Experimental): Drug: RN5681 Investigational product subcutaneous injections
  Interventions: Drug: RN5681
- Placebo (Placebo Comparator): Drug: Placebo control 0.9% normal saline subcutaneous injection
  Interventions: Drug: Placebo control

INTERVENTIONS:
Drug: RN5681 — Investigational Product
  Arms: RN5681
Drug: Placebo control — 0.9% normal saline SC injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and immunogenicity of single doses of RN5681 in Adult healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 18 to 35 kg/m2
* Fasting LDL-C ≥70 mg/dL (1.81 mmol/L) (all SAD cohorts); fasting LDL-C ≥100 mg/dL (2.59 mmol/L) (POC cohort only)
* Lp(a) at Screening: SAD cohort: ≥25 nmol/L POC cohort: ≥100 nmol/L
* Fasting triglycerides <400 mg/dL (4.51 mmol/L) at Screening
* No clinically significant abnormalities of hepatic or renal function

Exclusion Criteria:

* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >1.5× the upper limit of normal at screening
* Hemoglobin A1c (HbA1c) ≥6.5% at screening
* Current regular smoker (defined as >2 cigarettes/day or >10 cigarettes/week) within 3 months prior to screening
* Use of any siRNA, antisense oligonucleotide (ASO), cell and gene therapy, or clustered regularly interspaced short palindromic repeats (CRISPR) agent in the prior 12 months
* Received any prescription lipid-lowering medication, including but not limited to statins, ezetimibe, and PCSK9 inhibitors to alter serum lipids within 30 days before screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
in SAD cohort, To assess the safety and tolerability of subcutaneously (SC) administered RN5681 | From the enrollment to the end of treatment at Day180
  Incidence, severity, and causal relationship of adverse events (AEs) as reported by the Investigator, with severity determined according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v6.0
in POC cohort, To assess the metabolic markers of efficacy | From enrollment to the end of treatment at Day 180
  Percent change from Baseline in serum LDL-C and Lp(a) at Day 180

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Q-Pharm Pty Ltd., Brisbane, Queensland
  - Nucleus Network Pty Ltd., Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Undecided